CLINICAL TRIAL: NCT00934232
Title: A Phase I Open Label Study of IV Busulfan (Busulfex®) in Multiple Myeloma Patients 65 Years of Age or Older, or With Renal Insufficiency Undergoing Autologous Transplantation
Brief Title: Busulfan in Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Guido Tricot (Other)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Guido Tricot, Guido J.K. Tricot, MD, PhD, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32857
Record Dates: First submitted 2009-06-04; First posted 2009-07-08 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma
Keywords: cancer; myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Neoplasms, Plasma Cell | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Busulfan (Experimental): Busulfex given to patients who are either ≥65 years or have renal insufficiency
  Interventions: Drug: Busulfan

INTERVENTIONS:
Drug: Busulfan — Busulfan (Bu) is a bifunctional alkylating agent currently used almost exclusively as a component of conditioning regimens for both autologous and allogeneic stem-cell transplants.
  Other Names: Busulfex ®

SUMMARY:
Two main objectives of the study are:

Primary:

To determine the MTD of Busulfex ® that can be given safely over the least number of days to myeloma patients who are either ≥65 years of age (Group 1) or have renal insufficiency (Group 2), defined as creatinine >3mg/dL or creatinine clearance <30 mL/min.

Secondary:

To perform pharmacokinetic (PK) studies to evaluate individual variability and the relationship to toxicities in each of the two groups at each proposed dose level.

DETAILED DESCRIPTION:
This study is for first line treatment for multiple myeloma patients in patients >65 years or have renal insufficiency Busulfan introduces cytopenia much slower than melphalan while the time to recover after transplantation is the same. The duration of cytopenia with busulfan should therefore be shorter. Busulfan given in myeloma patients with renal failure has proven to be effective.

The initial proposed dose level in our study will be 3.2mg/kg of body weight over 6 hours for 3 days. The next levels will be 3.2mg/kg of body weight over 6 hours for 4 days, 4.3 mg/kg of body weight over 6 hours for 3 days, 5.6 mg/kg of body weight over 6 hours for 2 days, and 6.4 mg/kg of body weight over 6 hours for 2 days. Three patients per group will be entered at the first level. Further enrollment will be dependent upon toxicities observed. All dose escalations will be initiated after the PI has reviewed the toxicity data available on the prior dose levels and confirms that it is safe to proceed to subsequent dose level(s). Maximum tolerated dose will defined as the dose level immediately below the dose level at which ≥ 2 of 6 patients experiences a grade 4 non-hematological toxicity that is unexpected, related, and serious, and it will be evaluated separately for patients > 65 years of age or in patients with renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have ≥ 3 x 106 CD34 cell/kg in storage for this study.
2. Subjects must have symptomatic multiple myeloma at their new patient consult at HCI that, in the opinion of the enrolling physician, requires treatment.
3. Subjects must be at least 65 years of age and/or diagnosed with renal insufficiency, defined as serum creatinine ≥3mg/dL or a creatinine clearance of less than 30mL/minute.
4. Subjects must not have a history of chronic obstructive or chronic restrictive pulmonary disease. Subjects must demonstrate adequate pulmonary function studies defined as ≥50% of predicted on mechanical aspects (FEV1, FVC) and diffusion capacity (DLCO).
5. Subjects must demonstrate adequate cardiac function (≥40% LVEF on ECHO or MUGA).
6. Subjects must demonstrate adequate liver functions with total bilirubin and transaminase levels no higher than 1.5 times the institutional upper limit of normal. (If total bilirubin is > 1.5 times the upper limit of normal, a direct bilirubin needs to be assessed. Subject eligible as long as the direct bilirubin is not > 1.5 times the upper limit of normal)
7. Subjects must have at least one evaluable myeloma marker by which to judge response: serum M protein >1g/dL, free light chains in the serum that more than four times the upper limit of normal, urine M protein of ≥ 500 mg, urine free light chains of ≥ 500 mg/day, bone marrow plasmacytosis with >20% plasma cells, extramedullary plasmacytosis, or MRI/FDG-PET/CT scan demonstrating 1 or more focal lesions due to myeloma.
8. Subjects must have a SWOG performance score of 0-2 unless due to myeloma-related bone pain.
9. Subjects must be informed of the investigational nature of the study and must sign an IRB-approved informed consent in accordance with institutional and federal guidelines.
10. Female participants of child-bearing potential must have a negative pregnancy test documented within 10 days of enrollment.

Exclusion Criteria:

1. Subjects must not have serum transaminases >1.5 times the upper limit of normal and/or a direct bilirubin >1.5 time the institutional upper limit of normal (direct bilirubin to be assessed only if the total bilirubin is > 1.5 times the upper limit of normal)
2. Subjects must not be HIV positive or have active Hepatitis B or Hepatitis C infection. If serology antibody studies are positive, a quantitative PCR must be done to confirm.
3. Subjects must not have a prior malignancy in which life expectancy, which in the opinion of the investigator, is more likely to be determined by the prior malignancy than the myeloma. Patients must not be currently receiving therapy for the prior malignancy.
4. Subjects must not have had a prior autologous or allogeneic bone marrow transplant.
5. Subjects must not be pregnant or nursing. Women and men of reproductive potential may not participate unless they agree to use an effective contraceptive method.
6. Patients who have < 3 million CD34 cells/kg stored for this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
determine MTD of Busulfex given safely over least number of days patients who are either ≥65 years Group 1) or have renal insufficiency (Group 2), defined as creatinine >3mg/dL or creatinine clearance <30 mL/min. | 1 year

SECONDARY OUTCOMES:
To perform pharmacokinetic (PK) studies to evaluate individual variability and the relationship to toxicities in each of the two groups at each proposed dose level. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Guido Tricot, MD, PhD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: No